CLINICAL TRIAL: NCT07389863
Title: Evaluation of Gynecological and Sexual Sequelae in Patients Treated for Rectal Cancer
Brief Title: Evaluation of Gynecological and Sexual Sequelae
Acronym: GYNERECT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0441/OB; 2025-A02592-47 (Other: ANSM)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer Patients
Keywords: Gynecological and sexual sequelae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prevalence of gynecological and sexual sequelae in women after treatment for rectal cancer: The prevalence and characterization of gynecological and sexual sequelae in women after treatment for rectal cancer will be carried out on the basis of questionnaires under study (FSFI, QLQ-CR29, QLQ-C30 and the GynéRect questionnaire) completed during the single follow-up visit.

SUMMARY:
Rectal cancer accounts for approximately 40% of colorectal cancers. In France, there are 15,000 new cases per year, and the 5-year survival rate is 55% across all stages. Treatment involves surgical resection of the rectum, often combined with preoperative chemoradiotherapy and sometimes immunotherapy, depending on the tumor's immunohistochemical status.

This treatment strategy has improved recurrence-free survival but is associated with long-term functional complications affecting the digestive, urological, gynecological, and sexual systems. Surgery causes anatomical changes and damage to the autonomic nervous system plexuses. Radiotherapy, for its part, causes pelvic inflammation with the development of fibrosis and potential vascular and nerve damage.

Various disorders can arise as a result of these anatomical changes, such as erectile dysfunction in men; dyspareunia and vaginal dryness in women; urinary incontinence and impaired sexual quality of life in both sexes.

DETAILED DESCRIPTION:
In women, there is a significant link between gynecological clinical abnormalities and the onset of sexual dysfunction. Gynecological anatomical sequelae are a major determinant of female sexual health. However, their assessment in clinical practice in the context of rectal cancer remains inconsistent, incomplete, or delayed. The repercussions of impaired sexual quality of life are also significant from a public health perspective. Good sexual quality of life is directly linked to a better overall quality of life in women over 40. These results could therefore be extrapolated to patients experiencing sexual dysfunction after treatment for rectal cancer. Finally, impaired overall quality of life leads to increased healthcare utilization and disability, with significant socioeconomic repercussions.

Gynecological and sexual sequelae following treatment for rectal cancer are therefore frequent but insufficiently assessed and managed in clinical practice, despite their impact on patients' overall quality of life and on public health. This work would allow for a better understanding of these disorders in order to prevent, assess, and manage them more effectively and thus optimize patients' future quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 60 at the time of diagnosis
* Having been treated for rectal cancer between 2020 and 2025
* Cancer in remission
* Having been sexually active before receiving treatment for their rectal cancer
* Having completed the various questionnaires during their treatment

Exclusion Criteria:

* Inability to complete questionnaires (cognitive impairment, language barrier)
* Pregnant women
* Women with active cancer and/or undergoing chemotherapy
* Women with a history of extensive gynecological surgery
* Individuals deprived of their liberty by an administrative or judicial decision, or individuals under legal protection/guardianship or curatorship
* Individuals without social security coverage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing treatment for rectal cancer benefit from regular follow-up consultations with the digestive surgeon, allowing for the estimation of the prevalence and characteristics of sexual dysfunctions and gynecological sequelae through questionnaires.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of sexual dysfunctions and gynecological sequelae in women after treatment for rectal cancer. | 1 day
  Evaluation of the prevalence of sexual dysfunctions and gynecological sequelae after treatment in women for rectal cancer, assessed using a standardized questionnaire combining validated questionnaires (FSFI, QLQ-C30, QLQ-CR29) and a specific GynéRect module for phenotyping disorders
To assess the characteristics of sexual dysfunctions and gynecological sequelae in women after treatment for rectal cancer. | 1 day
  Evaluation of the description of sexual dysfunctions and gynecological sequelae after treatment in women for rectal cancer, assessed using a standardized questionnaire combining validated questionnaires (FSFI, QLQ-C30, QLQ-CR29) and a specific GynéRect module for phenotyping disorders

SECONDARY OUTCOMES:
Identify the main risk factors for gynecological and sexual sequelae in patients | 1 day
  The number of patients presenting the following risk factors will be assessed: menopausal status, treatment received (surgery alone, pre-operative radio-chemotherapy), surgical technique, tumor location, pelvic nerve involvement based on the medical data available in the computerized patient file and during questioning during a follow-up visit with the surgeon
Evaluate the relevance of the GynéRect questionnaire for assessing the gynecological and sexual sequelae of patients | 1 day
  However, to date, no validated questionnaire exists that allows for the precise and phenotypic assessment of sexual and gynecological sequelae after treatment for rectal cancer. For this reason, we propose the GynéRect questionnaire in this study.
Évaluer l'impact des séquelles gynécologiques et sexuelles des patientes sur leur qualité de vie globale | 1 day
  The criterion will be evaluated using the following questionnaires.The FSFI (Female Sexual Function Index) is an internationally validated self-administered questionnaire that assesses sexual function in women, including patients with a history of cancer. It consists of 19 questions evaluating six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Sexual dysfunction is defined as a score of 26.55 or higher on a scale of 36. Patients with an FSFI score ≥ 26.55 are therefore considered to have impaired sexual function.
  The QLQ-C30 questionnaire assesses health-related quality of life in cancer patients. It is an international standard and is recommended in most cancer clinical trials.
  The QLQ-CR29 questionnaire complements the QLQ-C30 by focusing on symptoms specifically related to rectal cancer, including bowel, urinary, and sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie VB BRIDOUX, Professor, Study Director — University Rouen Hospital; Pauline PL LUDWIG, Doctor junior, Principal Investigator — University Rouen Hospital
Locations (1):
- Service de Chirurgie Digestive, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.